CLINICAL TRIAL: NCT03719651
Title: Testing the Leadership and Organizational Change for Implementation (LOCI) Intervention in Norwegian Mental Health Clinics: A Stepped-wedge Design Study Protocol
Brief Title: Testing the LOCI Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: Principal Investigator, Karina Ester Myhren Egeland, Primary Investigator, Norwegian Center for Violence and Traumatic Stress Studies
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: LOCI Norway
Record Dates: First submitted 2018-07-05; First posted 2018-10-25 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Post-traumatic Stress Disorder; Leadership
Keywords: Implementation; Implementation strategy; Leadership; Organizational climate; Fidelity; PTSD treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Stepped wedge design with three cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): When clinics join the intervention arm, leaders will receive leadership training through the Leadership and Organizational Change for Implementation (LOCI) intervention.
  Therapists will receive training in evidence-based practices for treatment of Post-Traumatic Stress Symptoms (EMDR, CT-PTSD, TF-CBT)
  Interventions: Behavioral: LOCI; Behavioral: EMDR; Behavioral: CT-PTSD; Behavioral: TF-CBT
- Control (Active Comparator): Clinics that are not yet included in the intervention arm, the leaders will not receive any leadership training (LOCI).
  Therapists will receive training in evidence-based practices for treatment of Post-Traumatic Stress Symptoms (EMDR, CT-PTSD, TF-CBT)
  Interventions: Behavioral: EMDR; Behavioral: CT-PTSD; Behavioral: TF-CBT

INTERVENTIONS:
Behavioral: LOCI — LOCI includes training of leaders in general leadership, implementation leadership, and implementation climate.
  Arms: Intervention
Behavioral: EMDR — EMDR (Eye Movement and Desensitization Reprocessing), treatment method developed for treating patients with Post-Traumatic Stress Symptoms (PTSD).
Behavioral: CT-PTSD — CT-PTSD (Cognitive Therapy for PTSD), treatment method developed for treating patients with Post-Traumatic Stress Symptoms (PTSD).
Behavioral: TF-CBT — TF-CBT (Trauma-Focused Cognitive-Behavioral Treatment) treatment method developed for treating patients with Post-Traumatic Stress Symptoms (PTSD).

SUMMARY:
The project will develop knowledge on how managers can lead the implementation of practices that have proven to be effective for post-traumatic stress disorders (PTSD) in child and adult specialized mental health services. Specifically, the project will test the effectiveness of an intervention named the Leadership and Organizational Change for Implementation (LOCI). This is an empirically and theoretically based innovation for implementation leadership that aims to support leaders in their organizational work of leading the implementation of EBPs in their clinics.

It is hypothesized that the implementation of LOCI will improve leaders' general leadership qualifications, their implementation leadership qualifications, and the implementation climate in the clinics. Further, the investigators hypothesize that training in trauma screening will increase the amount of trauma screenings, moderated by the LOCI implementation, and also that training in trauma treatment will increase the amount of patients to be offered this kind of treatment, also moderated by the LOCI implementation.

DETAILED DESCRIPTION:
Leadership for implementation require leadership that supports effective implementation strategies at the organizational level. The Leadership and Organizational Change for Implementation (LOCI) is a leadership training program focusing on enhancing general leadership and implementation leadership in particular (Aarons, Ehrhart, Moullin, Torres, & Green, 2017). The aim of the project is to evaluate the implementation strategy used to implement evidence-based treatment for PTSD in child and adult specialized mental health services in Norway.

The Leadership and Organizational Change for Implementation (LOCI) consists of several components:

1. 360° assessment A 360° assessment where the LOCI leaders, the therapists who report to them, and the executive leader are asked to complete a web-based survey focused primarily on the leadership of the LOCI leader and the implementation climate in his/her unit. Questions to therapists and the executive leaders are worded so that they are reporting on the appropriate LOCI leader. The LOCI leaders are asked questions about their own leadership, climate in their clinic, and on the implementation citizenship of their therapists.

Descriptive results from the 360° assessment are presented in an individual feedback report for each of the LOCI leaders in the LOCI condition. Each of the LOCI leaders will receive their own feedback reports during the initial and follow-up leadership trainings, and they will not be required to share it with anyone besides the research group. Feedback reports for the executives will utilize data aggregated across all clinics within the respective health trusts. Executives will be presented with their feedback reports at initial and follow-up organizational strategy meetings (see below).

Leadership training 2.1 Training 2.1.1 Initial leadership training: The LOCI intervention begins with a two-day workshop for the LOCI leaders. The workshop addresses leadership in general, with a particular focus on the full-range leadership model, transactional leadership, and implementation leadership. The LOCI leaders are challenged to share own experiences and views on leadership, and examples of leadership styles are shared and discussed. Implementation climate is also addressed, with a focus on strategies leaders can use to support implementation of EBPs. Mid-way in the workshop at both day 1 and 2, the feedback reports from the 360° assessment will be shared individually with each of the LOCI leaders. The LOCI facilitator and the LOCI leader review the report together, identifying strengths and areas they would like to further develop. In a collaborative method, the LOCI facilitator and the LOCI leader draft that leader's individual leadership development plan wherein goals and committed actions are detailed to facilitate enhancement in their leadership and the implementation climate of their clinic.

2.1.2 Booster leadership training: The leadership training is followed by a one-day booster session after 4 and 8 months. Before each booster session, a new 360° assessment will be completed, resulting in updated feedback reports, where the data is presented in graphs so that it is easy to see the development from the baseline assessment to the assessment at 4 and 8 months. The feedback report makes the basis for the leaders´ subsequent work with the individual leadership development plan. Organizational strategies, goals, and leadership are addressed through group discussions.

2.1.3 Graduation: At month 12, there will be a ritual to mark the completion of the program. Accomplishments are celebrated, challenges are addressed, and plans for further sustainment are shared.

2.2 Coaching calls with first-level leaders The LOCI leaders will participate in weekly brief consultation calls over the phone (10-30 minutes) with their LOCI facilitator where the goals are to give the leaders the opportunities to strategize methods for overcoming barriers to EBP implementation; to follow up on the leadership development plan; and to update the leadership development plan according to the work being done and new information. Once a month the individual calls are replaced with one-hour group consultation calls with all the LOCI leaders within the cohort.

2.3 Organizational strategy meetings (OSMs) LOCI leaders and executives meet with the LOCI facilitator(s) for 2 hours following the first leadership training. The first meeting is in-person. At this meeting, the LOCI leaders and executives will receive feedback from the 360° survey followed by the iterative development of an implementation climate development plan in light of the results from the survey. The subsequent meetings take place on a web conferencing platform at months 4, 8, and 12. The executive will participate in brief (15-30 minutes) monthly telephone coaching calls with the LOCI facilitator where the focus is to follow up on the implementation climate development plan in light of the results from the 360° survey.

Evidence-based practices for post-traumatic stress disorders (PTSD) During the project, therapists will be trained in screening for and diagnosing PTSD, using evidence-based assessment tools. In addition, three well-documented EBPs for PTSD will be implemented in Norwegian specialized mental health services. 1) In child services, therapists will be trained in Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT) (Cohen, Mannarino & Deblinger, 2006). It builds on cognitive behavioral principle and incorporates principles from family therapy. In adult services, two practices will be implemented: 1) Eye Movement Desensitization and Reprocessing (EMDR) is an integrative eight-phase approach which is guided by the Adaptive Information Processing model (Shapiro & Laliotis, 2015). 2) Cognitive Therapy for PTSD (CT-PTSD) is based on a model assuming that PTSD develops if the traumatic event is processed in a way that maintains the experience of serious current threat (Ehlers & Clark, 2000).

Personnel in all clinics will receive training (2-3 hours) in screening for trauma and post-traumatic stress symptoms. A sample of therapists will receive three days of training in one of the specific practices (TF-CBT, EMDR, or CT-PTSD). In child services, the therapists will participate in 30 minutes weekly consultation group calls with 4-5 other TF-CBT therapists and a TF-CBT consultant. In adult services, the therapists will receive 10 hours of group consultation divided by 2 hours once a month for 5 months.

Methods:

A stepped wedge randomized trial will be used. The clinics will be allocated into three cohorts, based on which clinics to receive LOCI training at three different time-periods. The LOCI intervention lasts for 12 months. Allocation will be determined by an independent statistician. Co-located workgroups or closely working clinics will be assigned to the same condition to reduce the chances of contamination. The innovation effect is determined by comparing data points in the innovation section of the wedge with those in the control section.

The project will consist of three groups of participants:

1. First-level leaders will participate in the LOCI innovation and complete 360 degrees surveys. In addition, executive leaders will participate in organizational structural meetings to support first-level leaders, in addition to completing the surveys.
2. All therapists in the participating clinics will participate in the training of PTSD screening and the surveys. A sample of therapists will be trained and supervised in PTSD treatment.
3. Patients that are referred to the clinics as normal, report traumatic experiences and fulfill the criteria for PTSD will be offered to participate in the study. They will receive PTSD treatment, and complete surveys in connection with the treatment sessions.

The project aims at recruiting 20 child and youth mental health clinics and 20 adult mental health clinics in specialized services from all over Norway. The child and adult clinics will be recruited via the four regional health trust, which will receive an invitation by e-mail. Clinics may also receive information by the group giving lectures about the project in different settings.

Inclusion and exclusion criteria Child and adult outpatient clinics in specialized health services are included. All leaders and therapists in the clinics will be asked to participate in the surveys. Administrative personnel are excluded as most of the measures will not be applicable to these staff. Staff must be employees of the participating clinics. Leaders that do not agree to participate in the leadership training (LOCI) will not be eligible to participate.

Patients (6-100 years) with PTSD will be asked to participate in the study by their therapist. There are no specific exclusion criteria, as the referrals should follow standard procedures within the clinics.

Fidelity The TF-CBT therapists in the child clinics will audiotape all the trauma treatment sessions through an application on iPads specifically programmed for this project. Randomly chosen therapy sessions for each therapist will be checked for fidelity through a fidelity check list developed by the TF-CBT research group. Trained TF-CBT supervisors will do the fidelity assessments. The fidelity measure will be validated as part of this study. The therapists in the adult clinics will videotape (EMDR) or audiotape (CT-PTSD) all sessions in all cases. Randomly chosen therapy sessions for each therapist will be checked for fidelity. Students will be trained to assess five fidelity sessions per therapist. The therapists will receive written fidelity feedbacks as soon as possible after the session has been video or audiotaped.

Data collection and management Data are collected from therapists, LOCI-leaders, and executives from child and adult clinics at baseline, and at 4, 8, 12, 16, and 20 months. The surveys are distributed by e-mail. Participants are not given any compensation for their participation. The therapist and LOCI leader survey takes on average 25 minutes to complete, whereas the executive survey takes on average 15 minutes to complete. Results from some of the scales will be shared with the LOCI leaders (, MLQ, ILS, ICS, IC, EBPAS, ) and the executive leaders (ICS, IC, and EBPAS)) as part of the LOCI.

Patients will fill out a questionnaire by iPad in connection with all therapy sessions. It takes on average 30 minutes to complete. Patients can receive trauma treatment even if they do not want to participate in the research. All data will be stored on the University center for sensitive data and the Norwegian Centre for Research Data. Results from some of the scales will be shared with the therapist by a report function on the iPad.

Discussion Implementation of EBP can be challenging. Leaders in the health care system have the responsibility that the services provide effective treatments to a certain number of patients within a given time period. In order to increase the probability that patients will receive the most effective care for their symptoms, the leaders have to obtain effective strategies to promote the adoption of the evidence-based treatment. The LOCI intervention addresses leadership in general, implementation leadership in particular, and organizational strategies in order to support the implementation of EBP and sustainment over time. Available data suggest that LOCI is effective in supporting implementation of EBP through strengthening leadership and a positive implementation climate (Aarons et al., 2017). This study will examine the adaption of LOCI in a Norwegian mental health setting. A stepped wedge design will be used to investigate whether the LOCI will have an effect on leadership, the implementation climate at the clinics, and the clinic´s ability to offer trauma-focused treatments to patients with elaborated levels of post-traumatic stress symptoms. The knowledge derived from this study can be used to support the implementation of other EBPs within the mental health system.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary child and adult specialized mental health clinics that agree to the terms and conditions of the project, that is training, recruitment of patients, and data collection.
* Patients with PTSD symptoms and that agree to participate in the project.

Exclusion Criteria:

* Clinics or patients that do not agree to the terms and the conditions of the project

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Implementation Leadership Scale (ILS) | 4 weeks
  ILS assesses the degree to which leaders are knowledgeable, proactive, perseverant, and supportive during evidence-based practice (EBP) implementation.Scored from 0 (not at all) to 4 (to a very great extent).

SECONDARY OUTCOMES:
Number of trauma assessments and patients that receive trauma treatment. | 12 months
  Practitioners are asked to report the number of trauma assessments done within the last 4 months. The practitioners that have been trained in either TF-CBT, EMDR or CT-PTSD will also be asked to report the number of patients that receive the specific treatment.
The Multifactor Leadership Questionnaire (MLQ) | 12 months
  A 36-item measure addressing transformational and transactional leadership. Scored from 0 (not at all) to 4 (frequently, if not always)
The Implementation Climate Scale (ICS) | 12 months
  An 18-item measure addressing to what extent an organization support the implementation of EBP. Scored from 0 (not at all) to 4 (to a very great extent).
The Implementation Climate (IC) | 12 months
  A 6-item measure addressing the implementation climate in the organization. Scored from 0 (not at all) to 4 (often, if not always).
Workload (QPS) | 12 months
  Thirteen items from the QPS Nordic questionnaire. Coping with work (6 items), job demands (7 items). Scored from 1 (very seldom or never) to 5 (very often or always).
The Implementation Citizenship Behavior Scale (ICBS) | 12 months
  A six-item measure addressing employee behaviour that goes beyond their duty to support the implementation of EBP. Scored from 0 (Not at all) to 4 (Frequently, if not always).
TF-CBT Fidelity | 12 months
  Evaluating whether the therapist carries out the manual correctly. Developed for this Project.
The Treatment integrity checklist for EMDR (T-TIP EMDR) | 12 months
  consists of 16 items evaluating whether the therapist carries out the manual correctly ("yes" or "not relevant" = 1 point, "no" = 0 point). Maximal score is 16 points.
Cognitive Therapy for Post-Traumatic Stress Disorder: A Checklist of Therapist Competency | 12 months
  consists of 16 items evaluating therapists' general and specific therapeutic skills on a range between 0 (poor) and 6 (excellent)
The Child & Adolescent Trauma Screening Questionnaire (CATS) | 12 months
  20 symptom items and 5 functional impairment items. A total symptom severity scale score ranging from 0 to 60 is calculated. Screening cut off point is 15.
Stressful Life Events Screening Questionnaire - revised (SLESQ) | 12 months
  15 questions on stressful life events (0 = no, 1 = yes)
PTSD Checklist (PCL-5) | 12 months
  20 symptom items. A total symptom severity scale score ranging from 0 to 80. (0 = not at all, 4 = a lot)

CONTACTS AND LOCATIONS:
Overall Officials: Karina M Egeland, PhD, Principal Investigator — Norwegian Centre for Violence and Traumatic Stress Studies (NKVTS)
Locations (1):
- Karina Egeland, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egeland KM, Borge RH, Peters N, Baekkelund H, Braathu N, Sklar M, Aarons GA, Skar AS. Individual-level associations between implementation leadership, climate, and anticipated outcomes: a time-lagged mediation analysis. Implement Sci Commun. 2023 Jul 11;4(1):75. doi: 10.1186/s43058-023-00459-7. PMID 37434244
- [Derived] Skar AS, Braathu N, Peters N, Baekkelund H, Endsjo M, Babaii A, Borge RH, Wentzel-Larsen T, Ehrhart MG, Sklar M, Brown CH, Aarons GA, Egeland KM. A stepped-wedge randomized trial investigating the effect of the Leadership and Organizational Change for Implementation (LOCI) intervention on implementation and transformational leadership, and implementation climate. BMC Health Serv Res. 2022 Mar 4;22(1):298. doi: 10.1186/s12913-022-07539-9. PMID 35246135
- [Derived] Borge RH, Skar AS, Endsjo M, Egeland KM. Good soldiers in implementation: validation of the Implementation Citizenship Behavior Scale and its relation to implementation leadership and intentions to use evidence-based practices. Implement Sci Commun. 2021 Dec 11;2(1):136. doi: 10.1186/s43058-021-00240-8. PMID 34895347
- [Derived] Egeland KM, Skar AS, Endsjo M, Laukvik EH, Baekkelund H, Babaii A, Granly LB, Husebo GK, Borge RH, Ehrhart MG, Sklar M, Brown CH, Aarons GA. Testing the leadership and organizational change for implementation (LOCI) intervention in Norwegian mental health clinics: a stepped-wedge cluster randomized design study protocol. Implement Sci. 2019 Mar 13;14(1):28. doi: 10.1186/s13012-019-0873-7. PMID 30866973
- See also: Norwegian webpage for the implementation within adult mental health services — https://www.nkvts.no/prosjekt/implementering-av-traumebehandlingstilbud-til-voksne-itv/
- See also: Norwegian webpage for the implementation within child mental health services — https://www.nkvts.no/prosjekt/ledelse-og-implementering-av-tf-cbt/